CLINICAL TRIAL: NCT07350954
Title: Assessing the Acceptability and Feasibility of TRUST, a Brief Intervention for Paranoia in Adolescents.
Brief Title: Acceptability and Feasibility of a Brief Paranoia Intervention.
Acronym: TRUST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lucy Jonas (Other)
Responsible Party: Sponsor-Investigator, Lucy Jonas, Chief Investigator, Royal Holloway University
Organization: Royal Holloway University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RoyalHollowayTRUST
Record Dates: First submitted 2025-12-08; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Paranoia
Keywords: Paranoia; Adolescents; Child and Adolescent Mental Health Service; Feasibility; Acceptability; Mental Health
MeSH Terms: conditions — Paranoid Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TRUST (Experimental): A six-session individual psychological intervention combining values-based and mental imagery techniques for adolescents experiencing paranoia.
  Interventions: Behavioral: TRUST

INTERVENTIONS:
Behavioral: TRUST — Participants will receive TRUST, a six-session individual psychological intervention designed for adolescents who experience frequent or distressing suspicious thoughts about others. The intervention includes values-based work to identify what matters most to the young person, and mental imagery techniques aimed at modifying distressing beliefs about the self and others.
  Session 1: Assessment, Formulation and Psychoeducation Session 2: Values and value based goals Session 3-5: Harnessing imagery to pursue values and imagery focussed strategies to change negative beliefs about self and others Session 6: Bringing it all together and review.

SUMMARY:
The goal of this feasibility and acceptability trial is to test whether a new brief talking therapy can be successfully provided to and is suitable for adolescents (16-18) who are seeking help from Child and Adolescent Mental Health Services (CAMHS).

The main research question for the current study is: Is it feasible and acceptable to offer a brief values-based (helping young people identify what matters most to them) and imagery (using imagination to visualise positive experiences) intervention for adolescents experiencing paranoia in CAMHS?

It also aims to identify preliminary clinical outcomes, particularly changes in paranoia severity as measured by the Revised Green et al., Paranoid Thoughts Scale (R-GPTS).

Participants will complete an eligibility assessment and those eligible will be offered a six-session intervention. Assessment measures will be completed before, during and after the intervention.

DETAILED DESCRIPTION:
Paranoia involves intense fears that others intend to cause harm. This fear of being under threat and unable to trust others often causes a young person significant distress and impairs everyday functioning. Paranoia is common in adolescence (20-30% report weekly fears, rising to 35% among those seeking mental health care), occurring not only in psychosis but across a range of mental health disorders. Help-seeking adolescents with various non-psychotic conditions commonly report paranoid thoughts. Despite the prevalence and impact, there are currently no proven therapies designed specifically for young people experiencing paranoia. This trial aims to address this gap.

Current treatments for paranoia focus almost exclusively on adults. In adult populations, values-based approaches and mental imagery techniques have shown promise in reducing paranoia. These interventions address underlying cognitive processes, negative beliefs about self and others, distressing mental images, and lack of values-directed behaviour, which maintain paranoid thinking. However, youth mental health interventions require developmentally appropriate approaches.

This study's primary aim is to evaluate the feasibility and acceptability of delivering a brief psychological intervention to adolescents experiencing paranoia. Feasibility will assess whether the intervention can be practically delivered within a CAMHS setting, including recruitment capability, participant retention, and completion of study procedures. Acceptability will examine whether young people find the intervention suitable.

Secondary aims include exploring preliminary clinical outcomes. We will examine changes in paranoia symptoms, self and other beliefs, mental imagery, valued action and day-to-day functioning.

This study employs a single-case experimental design (SCED) with multiple baseline lengths (2, 3 and 4 weeks).

After screening for eligibility and completing pre-intervention questionnaires, participants begin a randomly assigned baseline phase to establish stable symptom measurement. Participants then receive six weekly one-hour individual therapy sessions. Outcome measures are completed throughout the intervention to track changes.

One month post-intervention, participants complete a follow-up assessment with the same outcome measures to evaluate maintenance of treatment effects and provide further feedback on their experience.

This feasibility trial addresses a critical treatment gap for adolescent paranoia. If successful, findings could guide the development of larger definitive trials. Positive findings could contribute to the development of evidence-based interventions for young people experiencing paranoia in routine mental health services.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16-18
* Seeking help from a Child and Adolescent Mental Health Service (CAMHS)
* A score ≥ 11 on the R-GPTS (Scale B)
* Sufficient understanding of English
* Capacity to consent, as assessed during the initial interview
* Wanting support with paranoia
* Low- moderate mental health risks (emotional difficulties that impact functioning, but no immediate risk to safety e.g., no suicidal intent).

Exclusion Criteria:

* Severe comorbid diagnoses apparent at the initial assessment (e.g., a primary alcohol or substance dependence issue measured using standardised assessments)
* The presence of a developmental disability or cognitive impairment that would interfere with participation.
* Concurrent participation in another psychological therapy
* High levels of current risk (e.g., significant and immediate concerns about the young person's safety, such as suicidal intent).

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Recruitment | From screening to completion of recruitment (up to 6 months)
  Recruitment looks at how many young people can be identified, screened, and enrolled into the study. This will show whether it is practical to recruit young people with paranoia from a CAMHS waiting list.
  GREEN: ≥ 5 participants of target recruited AMBER: 3 to 4 of target recruited RED: ≤ 2 of target recruited.
Retention | From enrolment to one-month follow-up (up to 14 weeks)
  Retention refers to how many participants stay in the study until the end. We will record how many young people complete all six therapy sessions and complete the end-of-therapy and one-month follow-up questionnaires. This shows whether young people are willing and able to stay involved in the study.
  GREEN: ≥5 participants providing end of therapy assessment outcome data AMBER: 3-4 participants providing end of therapy assessment outcome data RED: ≤2 participants providing end of therapy assessment outcome data
Adherence | From first therapy session to final therapy session (up to 6 weeks).
  Adherence describes how well participants follow the study schedule, including how many therapy sessions they attend.
  GREEN: ≥5 participants attend at least 3 sessions of therapy AMBER: 3-4 participants attend at least 3 sessions of therapy RED: ≤2 participants attend at least 3 sessions of therapy
Acceptability | Throughout the study, at the end of therapy, and at one month follow up (up to 14 weeks)
  Acceptability looks at how young people experience the intervention and whether they find it suitable and helpful. Acceptability of the therapy will be assessed via questionnaires given to participants upon therapy completion or withdrawal and adverse effects of study participation questionnaire.

SECONDARY OUTCOMES:
Paranoia - Revised Green et al., Paranoid Thoughts Scale (R-GPTS) Part B | Screening, before intervention (baseline), weekly baseline, each therapy session (weeks 1-6) and at one-month follow-up (up to 14 weeks).
  To screen for and measure paranoia, the study uses the R-GPTS. This questionnaire has 18 items split into two parts: 8 questions about ideas of reference and 10 questions about persecution (feeling that others intend to harm you). The study uses Part B (persecution subscale). Scores of 11 or higher on the persecution scale indicate clinically significant paranoid thoughts. Higher scores reflect greater difficulties with paranoia.
Negative Self and Other Beliefs - The Brief Core Schema Scales (BCSS) | Before intervention (baseline), after intervention (session 6; 6 weeks), and at one-month follow-up.
  Research has found that holding more negative views about oneself and others are linked to paranoia. The BCSS (Fowler et al., 2006) is a 24-item self-report measure assessing beliefs about the self and others using rating scale from zero (do not believe this) to four (believe it totally). It has strong internal consistency (α = .79 for positive-self and α = .84 for negative self) in clinical samples. For positive-other and negative-other schemas, the alphas were .88 in clinical samples. The BCSS has been demonstrated to be valid, quick and easy.
Mental Imagery Characteristics - The Negative Mental Imagery Questionnaire (MIQ-N) | Before intervention (baseline), after intervention (session 6; 6 weeks), and at one-month follow-up.
  Research has found that distressing mental images play an important role in maintaining paranoia.The MIQ-N measures characteristics of mental imagery. There are 16-items and four sub-scales: intrusiveness, realness, controllability and beliefs.Participants rate how true each of the statements is for them on a seven-point scale. Higher scores mean that these images are more frequent and distressing. The subscales show strong reliability (α= 0.84-0.90),
Values - Comprehensive Assessment of Acceptance and Commitment Therapy processes for Youth (compACT-Y; Morey et al., 2024). | Before intervention (baseline), after intervention (session 6; 6 weeks), and at one-month follow-up.
  Research has found that living in line with personal values may help reduce distress associated with paranoia. This study uses the 7 values-based questions from the compACT-Y. These items ask how much they feel able to act in ways that matter to them and live in line with their personal values. Participants rate each statement on a 7-point scale from 0 (not at all true) to 6 (completely true). Higher scores indicate greater engagement in valued action. This has been identified as a valid and reliable measure for young people.
Functioning - Work and Social Adjustment Scale for Youth (WSAS-Y) | Before intervention (baseline), after intervention (session 6; 6 weeks), and at one-month follow-up.
  Research has shown that paranoia can impact an adolescent's ability to engage in everyday activities. The WSAS-Y is a five-item self-report measure that evaluates functional impairment across key life domains including work/school and relationships with family/friends. Severity is assessed using an nine-point scale, with greater scores indicating greater impairment. The WSAS-Y has demonstrated good psychometric properties (e.g., internal consistency: α = 0.84) and is developmentally appropriate for adolescent populations.

CONTACTS AND LOCATIONS:
Locations (1):
- Westminster's Child and Adolescent Mental Health Service, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
We request optional consent to share fully anonymised data with other researchers to support future studies. If consent is not given, or if confidentiality cannot be fully protected, individual participant data will not be shared.

REFERENCES:
- [Background] Morey A, Samuel V, Lewis M, Williams M. Validation of the comprehensive assessment of acceptance and commitment therapy processes for youth: The CompACT-Y. JCPP Adv. 2024 Aug 11;5(2):e12271. doi: 10.1002/jcv2.12271. eCollection 2025 Jun. PMID 40519958
- [Background] Parker A, Kingston J. Evaluating a values-based intervention for adolescence with high nonclinical paranoia: A schools-based randomised control trial. Cogn Ther Res. 2022;46:620-8. doi: 10.1007/s10608-021-10278-6
- [Background] Yung AR, McGorry PD, Francey SM, Nelson B, Baker K, Phillips LJ, Berger G, Amminger GP. PACE: a specialised service for young people at risk of psychotic disorders. Med J Aust. 2007 Oct 1;187(S7):S43-6. doi: 10.5694/j.1326-5377.2007.tb01336.x. PMID 17908025
- [Background] Kingston J, Ellett L. Self-affirmation and nonclinical paranoia. J Behav Ther Exp Psychiatry. 2014 Dec;45(4):502-5. doi: 10.1016/j.jbtep.2014.07.004. Epub 2014 Jul 22. PMID 25090449
- [Background] Garety PA, Freeman D. The past and future of delusions research: from the inexplicable to the treatable. Br J Psychiatry. 2013 Nov;203(5):327-33. doi: 10.1192/bjp.bp.113.126953. PMID 24187067
- [Background] van Os J, Reininghaus U. Psychosis as a transdiagnostic and extended phenotype in the general population. World Psychiatry. 2016 Jun;15(2):118-24. doi: 10.1002/wps.20310. PMID 27265696
- [Background] Oaie FE, Bower JL, Steel C. The development of the Negative Mental Imagery Questionnaire (MIQ-N). Behav Cogn Psychother. 2025 Mar;53(1):17-29. doi: 10.1017/S1352465824000304. Epub 2024 Oct 18. PMID 39421888
- [Background] Jassi A, Lenhard F, Krebs G, Gumpert M, Jolstedt M, Andren P, Nord M, Aspvall K, Wahlund T, Volz C, Mataix-Cols D. The Work and Social Adjustment Scale, Youth and Parent Versions: Psychometric Evaluation of a Brief Measure of Functional Impairment in Young People. Child Psychiatry Hum Dev. 2020 Jun;51(3):453-460. doi: 10.1007/s10578-020-00956-z. PMID 32006302
- [Background] Freeman D, Loe BS, Kingdon D, Startup H, Molodynski A, Rosebrock L, Brown P, Sheaves B, Waite F, Bird JC. The revised Green et al., Paranoid Thoughts Scale (R-GPTS): psychometric properties, severity ranges, and clinical cut-offs. Psychol Med. 2021 Jan;51(2):244-253. doi: 10.1017/S0033291719003155. Epub 2019 Nov 20. PMID 31744588
- [Background] Taylor CDJ, Bee PE, Kelly J, Emsley R, Haddock G. iMAgery focused psychological therapy for persecutory delusions in PSychosis (iMAPS): a multiple baseline experimental case series. Behav Cogn Psychother. 2020 Sep;48(5):530-545. doi: 10.1017/S1352465820000168. Epub 2020 Apr 8. PMID 32264985

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-22): https://cdn.clinicaltrials.gov/large-docs/54/NCT07350954/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-22): https://cdn.clinicaltrials.gov/large-docs/54/NCT07350954/ICF_001.pdf